CLINICAL TRIAL: NCT02133677
Title: A Phase II, Open-label, Single-arm, Multi-center Pilot Study to Evaluate the Efficacy and Safety of Whole-brain Radiotherapy With Concomitant Temozolomide in Lung Cancer and Breast Cancer Patients With Brain Metastases
Brief Title: A Phase II Multi-center Pilot Study of Concurrent Temozolomide and Whole Brain Irradiation in Lung Cancer and Breast Cancer Patients With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-IRB-102072-F
Record Dates: First submitted 2014-02-05; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-02

CONDITIONS: Lung Cancer and Breast Cancer Patients With Brain Metastases
Keywords: lung cancer and breast cancer patients with brain metastases
MeSH Terms: conditions — Lung Neoplasms | interventions — Temozolomide

ARMS (1):
- temozolomide+WBRT (Experimental): temozolomide: TMZ 200 mg p.o. q.d. x 5 days per week x 3 weeks WBRT:30 Gy in 15 fractions (2 Gy per fraction, 5 fractions per week)
  Interventions: Drug: temozolomide 100mg

INTERVENTIONS:
Drug: temozolomide 100mg — WBRT: 30 Gy in 15 fractions (2 Gy per fraction, 5 fractions per week) CT: TMZ 200 mg p.o. q.d. x 5 days per week x 3 weeks
  Other Names: Tamos 100mg capsule

SUMMARY:
Brain metastasis (BM) is among the most feared complications in cancer because even small tumors may cause incapacitating neurologic symptoms. It is observed in more than 50% of patients with lung cancer and 15% to 25% of patients with breast cancer. Temozolomide (TMZ) is an oral alkylating agent that crosses blood-brain barrier (BBB). This pilot study aims to evaluate the efficacy, safety and tolerability of whole-brain radiotherapy (WBRT) plus concomitant TMZ in lung cancer and breast cancer patients with BM.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed lung cancer or breast cancer at primary site
* Patient with inoperable brain metastases
* Female or male, ≥ 20 and < 65 years of age
* Karnofsky performance status (KPS) ≥ 70%
* Life expectancy ≥ 12 weeks
* Adequate organ function
* Willing and able to provide a written informed consent

Exclusion Criteria:

* Female of childbearing potential* who is pregnant/lactating or planning to be pregnant
* Male whose partner is planning to be pregnant
* Inability to swallow
* Meningeal carcinomatosis
* History of hypersensitivity to iodinated contrast media, temozolomide or any component of the study drugs
* Prior use of temozolomide
* Use of systemic chemotherapy within 2 weeks prior to the initiation of study treatment
* Prior surgery, chemotherapy or radiotherapy for a brain neoplasm
* Current use of valproic acid
* Use of any investigational product within 4 weeks prior to the initiation of study treatment
* Patient with any condition or disease which is considered not suitable for this study by investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | assessments will be conducted between 10 to 14 weeks after the end of treatment, all subjects will be followed every 3 months since Month 6 until completion of study (12 months after the last patient is enrolled) or death, whichever comes first.
  To evaluate the objective response rate (ORR) of WBRT plus concomitant TMZ treatment in lung cancer and breast cancer patients with BM.

SECONDARY OUTCOMES:
Progression free survival (PFS) | assessments will be conducted between 10 to 14 weeks after the end of treatment, all subjects will be followed every 3 months since Month 6 until completion of study (12 months after the last patient is enrolled) or death, whichever comes first.
  Progression free survival (PFS), Overall survival (OS), Change from baseline in MMSE scores, Change from baseline in SF-36

OTHER OUTCOMES:
Safety | safety of study treatments will be assessed by physician at each return. The safety for individual subject will be followed till 2 weeks after EOT.
  1. Change in lab data
  2. Adverse event(s) (AE)
  3. Serious adverse event(s) (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Wei Shueng, MD, Principal Investigator — Chief, Department of Radiation Oncology
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan